CLINICAL TRIAL: NCT06559332
Title: Randomized Trial of Coronary Artery Disease Assessment Strategies in Patients With Severe Aortic Stenosis Undergoing Transcatheter Aortic Valve Implantation
Brief Title: Coronary Artery Disease Assessment Strategies in TAVI Patients
Acronym: CAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Clinical Trials Unit Bern (CTU) (Unknown); Schweizerische Herzstiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CAT Trial
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Transcatheter Aortic Valve Replacement; Coronary Artery Disease; Heart Disease Risk Factors
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical event adjudication committee will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk-based management strategy without invasive coronary angiography (Experimental): Patients will not undergo routine coronary angiography prior to TAVI. Statin treatment of at least moderate intensity is recommended.
  Interventions: Diagnostic Test: Risk-based CAD management
- Routine invasive coronary angiography (Other): Routine invasive coronary angiography prior to TAVI. Percutaneous coronary intervention (PCI) recommended for coronary diameter stenosis of ≥ 80% (visual angiographic assessment) in coronary segments with a reference vessel diameter of at least 2.5 mm. Timing of PCI at the operators' discretion.
  Interventions: Diagnostic Test: Invasive coronary angiography

INTERVENTIONS:
Diagnostic Test: Risk-based CAD management — Patients will not undergo routine coronary angiography prior to TAVI. Statin treatment of at least moderate intensity is recommended.
  Arms: Risk-based management strategy without invasive coronary angiography
Diagnostic Test: Invasive coronary angiography — Routine invasive coronary angiography prior to TAVI. PCI recommended for coronary diameter stenosis of ≥ 80% (visual angiographic assessment) in coronary segments with a reference vessel diameter of at least 2.5 mm. Timing of PCI at the operators' discretion.
  Arms: Routine invasive coronary angiography

SUMMARY:
Coronary artery disease (CAD) and aortic stenosis frequently coincide. Before valve intervention, invasive coronary angiography is routinely performed to assess coronary status.

As the impact of percutaneous revascularization on clinical outcomes beyond symptom improvement is subject to debate and treatment of aortic stenosis itself reduces ischemic burden and symptoms, the benefit/risk balance of routine invasive coronary angiography prior to transcatheter aortic valve implantation (TAVI) is unclear.

The CAT Trial aims to compare a non-invasive risk management strategy to routine invasive coronary angiography for the assessment of coronary artery disease in patients with severe, symptomatic aortic stenosis selected to undergo TAVI with respect to adverse clinical outcomes at 3 years (primary objective) and patient reported outcome measures (secondary objective).

ELIGIBILITY:
Inclusion:

• Severe aortic stenosis defined by aortic valve area (AVA) ≤1cm2 AND mean gradient ≥40 mmHg or peak velocity ≥4.0 m/s

OR

if mean gradient <40 mmHg and peak velocity (Vmax) <4 m/s and stroke volume indexed to body surface area (SVi) ≤ 35 mL/m2 and LVEF ≥50% then if CT-derived aortic valve calcium score >2000 Agatston units in men, >1200 in women

OR

if mean gradient <40 mmHg and Vmax <4 m/s and SVi ≤ 35 mL/m2 and LVEF <50% then if CT-derived aortic valve calcification >2000 Agatston units in men, >1200 in women OR if low-dose dobutamine stress echocardiography with flow reserve (>20% increase in stroke volume) and AVA ≤1cm2

* Coronary calcium score ≥ 400 Agatston units (derived from routine pre-TAVI CT) or known coronary artery disease
* Selected for treatment with transfemoral TAVI.
* Written informed consent.

Exclusion Criteria:

* Concomitant valvular heart disease or ascending aortic aneurysm with indication for surgery or intervention
* Unprotected left main coronary stenosis >50% or left main not evaluable based on coronary computed tomography angiography derived from routine pre-TAVI CT
* Left ventricular ejection fraction (LVEF) < 30%
* New regional wall motion abnormalities on echocardiography
* Myocardial infarction in previous 12 months
* Coronary angiography in previous 12 months
* Prior left main stenting

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death, myocardial infarction, any stroke, and heart failure hospitalization | 3 years
  Primary endpoint. Valve Academic Research Consortium (VARC)-3 definitions)

SECONDARY OUTCOMES:
Patient reported health status | 3 months, 1, 3 and 5 years
  Seattle Angina Questionnaire-7 (score from 0 to 100, with higher values indicating better health)
Patient reported health status | 3 months, 1, 3 and 5 years
  Kansas City Cardiomyopathy Questionnaire-12 (score from 0 to 100, with higher values indicating better health)
Patient reported health status | 3 months, 1, 3 and 5 years
  EuroQol 5D 5L (index scores range from -0.59 to 1, with higher values indicating better health)
Rate of all cause death | 3 months, 1, 3 and 5 years
Rate of cardiovascular death | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of disabling strokes | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of myocardial infarction | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of unplanned, urgent revascularization | 3 months, 1, 3 and 5 years
Rate of elective revascularization | 3 months, 1, 3 and 5 years
Rate of cardiovascular hospitalization | 3 months, 1, 3 and 5 years
Rate of heart failure hospitalization | 3 months, 1, 3 and 5 years
Rate of bleeding | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of acute kidney injury | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of tachyarrhythmia | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of major vascular complications | 3months, 1, 3 and 5 years
  (VARC-3)
Rate of major cardiac structural complications | 3 months, 1, 3 and 5 years
  (VARC-3)
Rate of permanent pacemaker implantation | 3 months, 1, 3 and 5 years
  (VARC-3)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Lanz, MD, MSc, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Department of Cardiology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
sharing via https://boris.unibe.ch platform
Supporting Information: Study Protocol, CSR
Time Frame: after study completion
Access Criteria: Data will be made available upon reasonable request